CLINICAL TRIAL: NCT02388841
Title: Assessment of the Association Between Thrombus Localization and Accompaying Disorders ,Rısk Factors, D-Dimer and Red Cells Distribution Witdh In Pulmonary Embolisim
Brief Title: Thrombus Localization and Accompaying Disorders and Risk Factors
Status: Completed | Type: Observational
Sponsor: Aysel Sünnetçioğlu (Other)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Sponsor-Investigator, Aysel Sünnetçioğlu, Department of Pulmory Diseas Aysel Sünnetçioğlu, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: YYU-015; YYU-2015-65 (Other: YUZUNCU YIL UNIVERSITY)
Record Dates: First submitted 2015-03-03; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism, Computed tomographic pulmonary
MeSH Terms: conditions — Pulmonary Embolism | interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pulmonary embolism: Distribution of the characteristics of Pulmonary Embolism patients according to thrombus localization
  Interventions: Radiation: Pulmonary embolism
- tomographic pulmonary angiography: Distribution of the characteristics of Pulmonary Embolism patients according to the localization of thrombi in the most proximal level of Main pulmonary artery and other arterial branches as confirmed by Computed tomographic pulmonary angiography
  Interventions: Radiation: Pulmonary embolism

INTERVENTIONS:
Radiation: Pulmonary embolism — the thrombus were assessed with Computed tomographic pulmonary angiography
  Other Names: Red cell distribution width

SUMMARY:
ABSTRACT Pulmonary embolism shows a wide spectrum ranging from clinically asymptomatic thrombus to massive thrombus, leading to cardiogenic shock. The purpose of this study was to determine the association between thrombus localization and risk factors, accompanying disorders, D-dimer and the red blood cell distribution width (RDW) in patients with pulmonary embolism.

DETAILED DESCRIPTION:
Background Pulmonary embolism shows a wide spectrum ranging from clinically asymptomatic thrombus to massive thrombus, leading to cardiogenic shock. The purpose of this study was to determine the association between thrombus localization and risk factors, accompanying disorders, D-dimer and the red blood cell distribution width (RDW) in patients with pulmonary embolism.

Material/Methods In 148 patients diagnosed with pulmonary embolism, the presence and anatomical localization of the thrombus were assessed with Computed tomographic pulmonary angiography. The accompanying disorders, risk factors, serum D-dimer, and the RDW in the patients were retrospectively evaluated.

Background Pulmonary embolism (PE) is a serious cardiopulmonary disorder caused by partial or complete obstruction of the pulmonary arterial bed by a thrombus formed in systemic veins. Pulmonary embolism is thought to be a result of the interaction between the patient and risk factors 1-3. In case of suspected PE, clinical, laboratory, and radiological findings should be carefully studied. Since the clinical findings in PE are non-specific, objective diagnostic tests are required for the diagnosis 4. Computed tomographic pulmonary angiography (CTPA) is increasingly being used as the first investigation for suspected PE. The extent of PE is commonly expressed by indicating the anatomical level of the most proximal vessel affected by a thrombus 5. For the definite diagnosis of suspected PE, one of the tests to be used is the determination of the D-dimer level. Plasma D-dimer measurement provides information about fibrin-degradation fragment following fibrinolysis. D-dimer assays have low specificity, but high sensitivity and negative predictive value in most patients with suspected thromboembolism 6. The red cell distribution width (RDW) is a quantitative indicator of the size variability of red blood cells. This parameter can be easily obtained from a full blood count and is accepted as an indicator of ineffective red cell production 7. Some studies have suggested that RDW may be associated with cardiovascular and pulmonary diseases including PE 8-13.

The purpose of this study was to determine the association between thrombus localization and risk factors, accompanying disorders, D-dimer and red blood cell distribution width (RDW) in patients with pulmonary embolism.

Material and Methods Study design The data confirmed on 148 patients having PE by CTPA in the Clinic of Chest Diseases, Medical School, Yüzüncü Yıl University, Van, Turkey, in the period between January 2012 and August 2014 were retrospectively studied. The patients' accompanying disorders, risk factors, and the dosing of D-dimer performed on the same day of the CTPA and RDW levels were noted. The patients who had a story of hospitalising for reasons other than surgery such as Pneumonia, apses, brucella, encephalitis and the bedridden patients such as hemiplegia and long-term immobilised patients (>72 hours) after surgery were listed in the immobilisation group.

Patients receiving the diagnosis of PE with no CTPA performed and 6 patients whose haemoglobin values were below 11 were not included in this study.

Computed tomographic pulmonary angiography A thoracic CT scan was performed using a 16-detector multi-sectional CT scanner (Somatom Emotion 16-slice; CT2012E-Siemens AG, Berlin and München-Germany) by injecting contrast agents intravenously, while the patient held her breath. Contrast-enhanced images were obtained 50-70 sec after IV administration of 120 ml of ionic iodinated contrast agent, iodiksanol (Visipaque 320 mg/100 ml, Opakim) using a power injector at a rate of 2 ml/sec.

The parameters used were 120-130 (Kv), 80-120 (Ef-Mass), 0.6 sec (rotation time), 16 mm×1.2 mm (acquisition), 1.2 mm (slice collimation), 5.0-3.0 (slice width), 0.80 (pitch factor), 5.0 mm (increment), and 512×512 (matrix).

D-dimer test The patients' blood specimens were evaluated in the Clinical Hematology Laboratory. The D-dimer levels were measured with a latex-enhanced photometric method ( Sta compact, Dade Behring, Marburg, Germany) using D-dimer kits.

Red blood cell distribution width (RDW) The red cell distribution width (RDW) was determined in whole blood specimens. The hematological analysis was performed with a Coulter LH 750 Complete Blood Count device (Beckman Coulter, Fullerton, California, USA).

The study was planned according to the Declaration of Helsinki and rules of the Hospital Ethics Committee.

Statistical analysis Descriptive statistics were presented with frequency and percent for categorical data, and with mean and standard deviation for numerical data. Comparisons between 2 independent groups were conducted with Mann-Whitney U test, and Chi-Square test for non-normally distributed numerical, and categorical variables, respectively. Pairwise Pearson correlation was executed to estimate linear relationship between characteristics. Receiver operating characteristic (ROC) curve analysis was utilized to determine the optimum cutoff level of the association of RDW with MPA. All statistical calculations were performed using SAS version 9.3 (SAS, 2014). The results were considered statistically significant when the p value was <0.05.

ELIGIBILITY:
Inclusion Criteria:

- Pulmonary embolism Computed tomographic pulmonary angiography Red cell distribution width

Exclusion Criteria:

- Patients receiving the diagnosis of PE with no CTPA performed and 6 patients whose haemoglobin values were below 11 were not included in this study.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data confirmed on 148 patients having PE by CTPA in the Clinic of Chest Diseases, Medical School, Yüzüncü Yıl University, Van, Turkey, in the period between January 2012 and August 2014 were retrospectively studied. The patients' accompanying disorders, risk factors, and the dosing of D-dimer performed on the same day of the CTPA and RDW levels were noted. The patients who had a story of hospitalising for reasons other than surgery such as Pneumonia, apses, brucella, encephalitis and the bedridden patients such as hemiplegia and long-term immobilised patients (>72 hours) after surgery were listed in the immobilisation group.
  Patients receiving the diagnosis of PE with no CTPA performed and 6 patients whose haemoglobin values were below 11 were not included in this study.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
association between thrombus localization and risk factors, accompanying disorders, D-dimer and red blood cell distribution width (RDW) in patients with pulmonary embolism. | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: aysel sunnetcioglu, PHD, Study Director — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University Hospital, Van, Tuşba, Turkey (Türkiye)

REFERENCES:
- [Derived] Sunnetcioglu A, Sertogullarindan B, Ozbay B, Asker S, Ekin S. Assessments of the associations of thrombus localization with accompanying disorders, risk factors, D-dimer levels, and the red cell distribution width in pulmonary embolism. Clinics (Sao Paulo). 2015 Jun;70(6):441-5. doi: 10.6061/clinics/2015(06)10. Epub 2015 Jun 1. PMID 26106964